CLINICAL TRIAL: NCT05528250
Title: The Effect of Quadriceps Muscle Fatigue on Static and Dynamic Balance in Regular Physical Activity and Sedentary Individuals
Brief Title: The Effect of Quadriceps Muscle Fatigue on Balance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Meryem Özdemir, Phsiotherapy Student, Saglik Bilimleri Universitesi
Other Study IDs: Balance and The Quadriceps
Record Dates: First submitted 2022-08-19; First posted 2022-09-06 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-08

CONDITIONS: Muscle Fatigue
Keywords: Quadriceps Muscle Fatigue; Static Balance; Dinamic Balance; Regular Physical Activity; Sedentary
MeSH Terms: conditions — Sedentary Behavior | interventions — Surveys and Questionnaires; Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- İndividuals with do regular physical activity: International Physical Activity Questionnaire (IPAQ)-Short Form ,Anthropometric Measurements and Evaluation Body Weight and Height, Electromyogram (EMG), Digital Dynamometer measurement ,Static Balance Measurements ,Dynamic Balance Measurements ,Tecnobody Balance Measurement , Mini-Balance Evaluation (MiniBESTest) Systems Test ,Y Balance Test ,Flamingo Balance Test ,Modified Borg Scale will be applied to individuals with do regular physical activity is declared.
  Interventions: Other: Survey; Device: Treadmill
- Sedentary individuals with do not have regular physical activity: International Physical Activity Questionnaire (IPAQ)-Short Form ,Anthropometric Measurements and Evaluation Body Weight and Height, Electromyogram (EMG), Digital Dynamometer measurement ,Static Balance Measurements ,Dynamic Balance Measurements ,Tecnobody Balance Measurement , Mini-Balance Evaluation (MiniBESTest) Systems Test ,Y Balance Test ,Flamingo Balance Test ,Modified Borg Scale will be applied to sedentary individuals with do not have regular physical activity is declared.
  Interventions: Other: Survey; Device: Treadmill

INTERVENTIONS:
Other: Survey — International Physical Activity Questionnaire (IPAQ)-Short Form ,Anthropometric Measurements and Evaluation Body Weight and Height, Electromyogram (EMG), Digital Dynamometer measurement ,Static Balance Measurements ,Dynamic Balance Measurements ,Tecnobody Balance Measurement , Mini-Balance Evaluation (MiniBESTest) Systems Test ,Y Balance Test ,Flamingo Balance Test ,Modified Borg Scale.
Device: Treadmill — Participants will sign a consent form approved by the ethics committee.Before data collection, height, weight, circumference measurements, leg length, thigh area subcutaneous fat measurement, heart rate, blood pressure and saturation values will be recorded. Before the muscle fatigue protocol, the muscle strength, balance assessment and fatigue of the participants will be evaluated. The muscle fatigue protocol will be done with a treadmill. At the end of the muscle fatigue protocol, the necessary evaluations will be made again and the participants will be rested.

SUMMARY:
This study; will be conducted to investigate the effect of quadriceps muscle fatigue on static and dynamic balance in regular physical activity individuals and sedentary individuals. International Physical Activity Questionnaire Short Form (IPAQ), Mini BESTest, Modified Borg Scale questionnaire and acute muscle fatigue protocol will be applied and Y balance Test, Flamingo Balance Test, Tecnobody Balance Measurement, EMG measurement, anthropometric measurements and digital dynamometer measurements will be made.

DETAILED DESCRIPTION:
Determining the dynamic or static balance of the person will enable us to determine the effect of physical activity levels on the balance in relation to muscle strength and provide us with information about the balance of the person and will give us workable data. Through to these data, we get information about whether the person's level of physical activity is at the desired level. If not, the exercises to be done to reach the desired level or the way the rehabilitation processes to be applied give us important clues in terms of choosing the methods to be applied and determining the direction in which the order will be. If the balance of the person is at the desired level, these data provide us with a great deal of convenience and guide the preservation of this balance.

Knowing the balance data in line with the results to be obtained with this study and using the tests or devices designed in this direction will increase the success of the rehabilitation process and constitute the most important part of the performance increase in physical activity levels.

In case of successful completion of the project, sedentary participants will turn to physical activity to increase their balance. Participants will reduce the risk of falling by increasing their balance by doing physical activity. Therefore, our study will be conducted to investigate the effect of quadriceps muscle fatigue on static and dynamic balance in regular physical activity individuals and sedentary individuals.

Following the approval off the ethics committee, a study will be conducted with 32 regular physical activity individuals and 32 sedentary individuals. The study will start with the approval of the ethics committee and is planned to be completed in May 2022, within 4 months.

Individuals who meet the inclusion criteria and voluntarily accepted to participate in the study will be administered the International Physical Activity Questionnaire Short Form (IPAQ), Mini BESTest, Modified Borg Scale questionnaire and acute muscle fatigue protocol will be applied and Y balance Test, Flamingo Balance Test, Tecnobody Balance Measurement, EMG measurement, anthropometric measurements and digital dynamometer measurements will be made to both regular physical activity individuals and sedentary individuals.

ELIGIBILITY:
Inclusion Criteria:

* Participant between the ages of 18-25.
* Participant volunteer for research.
* Have not had any lower extremity surgery.
* Not having any lower extremity injury in the last 6 months.
* Not having any chronic lower extremity pain.

Exclusion Criteria:

* People with chronic illness.
* Chronic diseases.
* Neurological problems.
* Cardiopulmonary problems.
* Cardiovaskular problems.
* Those who had any lower extremity injury during the study period.
* Being reluctant to continue research.

Ages: 18 Years to 25 Years | Sex: All
Age Groups: Adult
Study Population: Volunteers between the ages of 18-25 who do regular physical activity and are sedentary.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Superficial Electromyographic(EMG) Measurement | Change from baseline emg values in 30 minutes
  In the dominant lower extremity to evaluate muscle activity, vastus medialis and vastus lateralis, surface EMG signals will be recorded with the Trigno Avanti Wireless Surface EMG System. While the participant is standing in hip neutral and knee extension, the adhesive EMG electrode will be placed on the reference motor point. Superficial EMG values will be recorded throughout the exercise. During the research, EMG will be recorded from the stimulated muscles by applying two electrodes to the skin for each muscle. The amplitude, duration and shape of the evoked muscle action potentials obtained will be reflected as a result. The amplitudes of the EMG signals will be evaluated. The method to be used when evaluating EMG signal amplitudes will be the raw EMG calculation. While evaluating the data, the computer package programs will benefit.
Static-Dynamic Balance Evaluation with Isokinetic Balance Device | Change from baseline static and dynamic balance values in 30 minutes
  Static and dynamic balance performances will be evaluated using the isokinetic balance measurement system. In this system, there is a sensor in the center of the platform that detects every angular movement and sends the information directly to the computer. For the static balance test, it will be ensured that they stand on both feet with their eyes open. The arms will be positioned next to the body. The measurement will be recorded by asking the participants to maintain their stable position for 30 seconds. For the dynamic balance test, the difficulty level of the test will be set to "30". In the test, they will be asked to circle clockwise 5 times in 60 seconds without bending their knees within the limited area on the computer screen. The Patient Record database module enables the creation of clinical cards for each case. It facilitates the comparison of each case's own tests.
Static Balance | Baseline
  The flamingo balance test will be used to measure the static balance of the participants. Participants will be asked to stand on the 50 cm long, 3 cm wide and 4 cm high apparatus and balance for 1 minute. Every mistake of the participants when their balance is broken will be recorded as points.
Dynamic Balance | Baseline
  Y balance test will be used for the dynamic balance measurement of the participants. Participants will be asked to lie on the Y-shaped mechanism and lie in 3 directions. At least 3 stretches will be made in each direction and the amount of stretching will be recorded in cm.

SECONDARY OUTCOMES:
Evaluation of Leg Fatigue with the Modified Borg Scale (MBS) | Change from baseline muscle fatigue scale values in 30 minutes
  This scale was developed by Borg in 1970 to measure the effort expended during physical exercise. It is a scale that is frequently used to evaluate the severity of dyspnea on exertion and the severity of dyspnea at rest. It consists of ten items describing the severity of dyspnea according to their degrees. Defining the severity of dyspnea on the scale makes it easier for patients to apply. In the studies carried out; It is stated that MBS is a reliable scale for determining the severity of dyspnea at rest and exertion, and is associated with respiratory rate and pulmonary function tests. In addition, it is emphasized that MBS is superior to other scales in terms of long-term reproducibility and can be used to predict ventilatory reserves of patients.
Muscle Strength | Baseline
  Muscle strength measurement will be made with a digital muscle strength device.

CONTACTS AND LOCATIONS:
Overall Officials: Esra PEHLİVAN, assoc.prof, Study Director — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Istanbul, Kadıköy, Turkey (Türkiye)